CLINICAL TRIAL: NCT07143825
Title: A National Multicenter Epidemiological Investigation of Small Vulnerable Newborns in China
Brief Title: A National Multicenter Survey on Small Vulnerable Newborns
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-25-006
Record Dates: First submitted 2025-08-12; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Preterm; Small Gestational Age (SGA)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this nationwide multicenter observational study is to comprehensively investigate the severity of Small Vulnerable Newborns (SVN) issues across China and to propose further preventive and intervention measures. The primary aim is to provide a thorough description of SVN problems using a unified definition and framework, and to develop targeted prevention strategies.

Participating centers across the country will collect clinical data on vulnerable newborns under their care and complete detailed questionnaires to support this research.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns diagnosed as vulnerable infants at the participating hospitals between January 1 and December 31, 2024;
2. Meeting any one of the following criteria:

   * Diagnosed as small for gestational age (SGA): birth weight below the 10th percentile for infants of the same gestational age and sex;
   * Preterm infants: gestational age less than 37 weeks;
   * Low Birth Weight (LBW) infants: birth weight less than 2,500 grams.

Exclusion Criteria:

* Incomplete medical records due to missing data preventing comprehensive case evaluation.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Small vulnerable newborns admitted to major hospitals across various regions of China in 2024
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of small vulnerable newborns | From date of hospital admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 year.
Mortality rate | From date of hospital admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 year.

SECONDARY OUTCOMES:
Incidence of complications in small vulnerable newborns | From date of hospital admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 year.
  Including mechanical ventilation, bronchopulmonary dysplasia, congenital heart defects, congenital gastrointestinal malformations, retinopathy of prematurity, periventricular-intraventricular hemorrhage, periventricular leukomalacia, neonatal sepsis, and neonatal bacterial meningitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China